CLINICAL TRIAL: NCT06234579
Title: "GALILEO (Genomic ALteratIons and cLonal EvOlution in ALK+ NSCLC) - Valutazione Longitudinale Delle Alterazioni Genomiche e Clonali Nei Pazienti Affetti da Neoplasie Polmonari ALK-riarrangiate".
Brief Title: Longitudinal Assessment of Genomic Alterations and Clonal Evolution in ALK-positive NSCLC (Galileo Project)
Acronym: GALILEO
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Bria Emilio, Prof., Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 4906
Record Dates: First submitted 2023-04-10; First posted 2024-01-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: ALK Gene Mutation; NSCLC Stage IV; ALK Sensitizing Mutation
Keywords: ALK mutation; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Biopsy; Histocompatibility Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — At the time of diagnosis, all newly diagnosed ALK+ NSCLC patients eligible for first line treatment with alectinib or brigatinib or lorlatinib will be considered for the study.
  In case of progression, a multidisciplinary team (oncologists, interventional pneumologists and radiologists, surgeons) will discuss case-by-case the feasibility to procure an adequate biopsy from progressing lesions. Repeat biopsies will be performed within 2 weeks from multidisciplinary evaluation and before the start of subsequent treatment. If repeat biopsies are not technically or safely feasible or fail to yield sufficient material for genomic analysis, we will collect a whole blood drawn by venepuncture for the analysis of ctDNA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ALK+ NSCLC: The GALILEO project is an Italian observational prospective cohort study on advanced ALK+ NSCLC patient progressing on first-line therapy with alectinib
  Interventions: Diagnostic Test: Biopsy (tissue or liquid)

INTERVENTIONS:
Diagnostic Test: Biopsy (tissue or liquid) — At the time of diagnosis, all newly diagnosed ALK+ NSCLC patients eligible for first line treatment with alectinib or brigatinib or lorlatinib will be considered for the study.
  In case of progression, a multidisciplinary team (oncologists, interventional pneumologists and radiologists, surgeons) will discuss case-by-case the feasibility to procure an adequate biopsy from progressing lesions. Repeat biopsies will be performed within 2 weeks from multidisciplinary evaluation and before the start of subsequent treatment. If repeat biopsies are not technically or safely feasible or fail to yield sufficient material for genomic analysis, we will collect a whole blood drawn by venepuncture for the analysis of ctDNA.
  Other Names: Alectinib; Brigatinib; Lorlatinib

SUMMARY:
The scope of GALILEO project (Genomic ALteratIons and cLonal EvOlution in ALK+ NSCLC) is to explore the feasibility of genomic longitudinal evaluation for ALK+ NSCLC patients in Italian routine practice and provide a detailed overview of resistance mechanisms and clinical outcomes according to current standard treatments.

ELIGIBILITY:
Inclusion Criteria:

* a) histologically confirmed diagnosis of advanced NSCLC with ALK rearrangement detection by NGS (ALK+ NSCLCs patients detected at diagnosis by in hybridization (FISH), immunohistochememistry (IHC), or reverse transcriptase-PCR (RT-PCR) can be included if adequate tissue for NGS is available)

  b) to have received upfront treatment with alectinib, brigatinib or lorlatinib for at least 28 days

  c) ECOG PS 0-2

  d) adult patients (aged ≥ 18 years) at the moment of diagnosis

  e) signing of informed consent approved by the local Ethic Committee

Exclusion Criteria:

a) Diagnosis of lung cancer without ALK rearrangement

a) early withdrawn of treatment due to toxicity without evidence of radiological disease progression cannot be eligible for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed ALK+ NSCLC who are candidate to receive first-line therapy with II-III genaration ALK-inhibitor (alectinib, brigatinib or lorlatinib)
Sampling Method: Non-Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2021-07-12 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with available NGS testing at diagnosis | 5 years
  Percentage of ALK+ patients with adeguate tissue for NGS after diagnosisc biopsy
Percentage of patients with available NGS re-testing after progession (either tissue or ctDNA) to first-line treatment with II-III generation ALK-Inhibitor | 5 years
  Percentage of patients who obtenied successfull NGS post-progression testing after re-biopsy or liquid biopsy

SECONDARY OUTCOMES:
PFS to first-line treatment with II-III generation ALK-inhibitor | 5 years
  Time from treatment start until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years
PFS to first-line treatment with II-III generation ALK-inhibitor | 5 years
  Time from treatment start to death for any cause, assesed up to 5 years

OTHER OUTCOMES:
PFS to first-line treatment with II-III generation ALK-inhibitor | Time from treatment start until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years
  PFS to first-line, stratified according to ALK-rearrangement variants
PFS to first-line treatment with II-III generation ALK-inhibitor | Time from treatment start until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years
  PFS to first-line, stratified according to NGS-based mutational profiling
OS to first-line treatment with II-III generation ALK-inhibitor | Time from treatment start until the date of death from any cause, assessed up to 5 years
  OS to first-line, stratified according to ALK-rearrangement variants
OS to first-line treatment with II-III generation ALK-inhibitor | Time from treatment start until the date of death from any cause, assessed up to 5 years
  OS to first-line, stratified according to NGS-based mutation profiling
Incidence of secondary resistance mutations (SNVs) after first line treatment | 5 years
  Percentage of patients with SNV-based resistance diagnosed by tissue or liquid biopsy
PFS to lorlatinib according to secondary resistance mechanism | Time from treatment start until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years
  PFS to second-line lorlatinib, stratified according to type of resistance (SNV vs off-target)

CONTACTS AND LOCATIONS:
Overall Officials: GIAMPAOLO TORTORA, Prof., Principal Investigator — Fondazione Policlinico Universitario A Gemelli
Locations (1):
- Fondazione Policlinico Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No